CLINICAL TRIAL: NCT01170624
Title: Clinical Status Monitoring in ICD Patients by Physiological Diagnosis (PhD) Function
Brief Title: Clinical Status Monitoring in Implantable Cardiac Defibrillator (ICD) Patients by Physiological Diagnosis (PhD) Function
Acronym: TUTOR
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Field Safety Notice related to potential ventricular oversensing associated to the PhD feature on Paradym ICDs
Sponsor: LivaNova (Industry)
Responsible Party: Clinical Status Monitoring in ICD Patients by PhD functions, Sorin Group
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: TUTOR - ITSY04
Record Dates: First submitted 2010-06-16; First posted 2010-07-27 (Estimated); Last update posted 2015-01-12 (Estimated); Status verified 2015-01

CONDITIONS: Heart Failure
Keywords: PhD; EGM; CRT-D; The study will particularly focus on a new-based diagnostic feature, called PhD-Clinical Status (PhD)
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Device: ICD — Paradym CRT model 8750 - Paradym DR model 8550 - Paradym VR model 8250

SUMMARY:
The purpose of this study is to evaluate the performance of advanced features, that have been implemented in the PARADYM ICD Platform offering single chamber (VR - model 8250), dual Chamber (DR - 8550) and Cardiac Resynchronization System with defibrillation capabilities (PARADYM CRT System, model 8750) in a general ICD population.

DETAILED DESCRIPTION:
The study will particularly focus on a new sensor-based diagnostic feature, called PhD-Clinical Status (PhD). A dedicated PhD screen shows the trends of patients' ventilation levels at rest (MVR) and under effort (MVE), and the corresponding level of activity, day-by-day, over a period of 6 months.

ELIGIBILITY:
Inclusion Criteria:

1. Patient eligible for implantation of an ICD or a CRT-D device according to current available guidelines.
2. Documented chronic HF (NYHA Class II to IV) at the time of enrollment
3. Scheduled for implant of a PARADYM ICD / CRT-D or implanted within the previous month
4. Signed and dated informed consent

Exclusion Criteria:

1. Any contraindication for ICD therapy
2. Abdominal implantation site
3. Acute myocarditis
4. Unstable coronary symptoms (unstable angina or myocardial infarction) within the last month
5. Planned heart transplant
6. Mechanical tricuspid valve
7. Unable to perform the 6 minute Walking Test at time of enrollment
8. Already included in another clinical study
9. Life expectancy less than 13 months
10. Inability to understand the purpose of the study or refusal to cooperate
11. Inability or refusal to provide informed consent
12. Under guardianship
13. Age of less than 18 years
14. Pregnancy (Women of childbearing potential should have a negative pregnancy test prior to enrollment)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 388 (Actual)
Dates: Start 2009-09; Primary Completion 2011-09 (Actual); Study Completion 2011-09 (Actual)

PRIMARY OUTCOMES:
The objective is to demonstrate that agreement correlation is superior to 67% | 13 months

CONTACTS AND LOCATIONS:
Locations (25):
- Algemeen Ziekenhuis Middelheim Lindendref 1 2020 Antwerpen, Antwerp, Belgium
- France (14):
  - Centre Hospitalier Général, Albi
  - Centre Hospitalier Universitaire D'Amiens, Amiens
  - Chu Annecy, Annecy
  - CENTRE HOSP. HENRI DUFFAUT - Service de Cardiologie AVIGNON, Avignon
  - Hopital D'Instruction Des Armees, Clamart
  - Hôpital St Joseph, Lyon
  - Centre Hospitalier Universitaire de La Timone, Marseille
  - Hopital Le Raincy Montfermeil, Montfermeil
  - HOPITAL ARNAUD DE VILLENEUVE - Service de Cardiologie, Montpellier
  - Hopital de La Source, Orléans
  - Centre Hospitalier, Pau
  - CLINIQUE ST PIERRE Cardiologie, Perpignan
  - Ccn: Centre Cardiologique Du Nord St Denis, Saint-Denis
  - Chru Hôpital Trousseau, Tours
- Germany (5):
  - Kerckhoff Klinik Cardiology Department, Bad Nauheim
  - Lerckhoff Klinik, Bad Neuheim
  - Praxis Westend Studien GbR, Medianzentrum Haus 9, Berlin
  - Klinik Frankische Schweiz, Ebermannstadt
  - Med. Univ. Klinik Lübeck, Lübeck
- Italy (2):
  - Spedali Civili Divisione di Cardiologia, Brescia
  - Azienda Ospedaliera S. Croce E Carle, Cuneo
- Portugal (3):
  - Hospital de Santa Cruz - Carnaxide (Adragão), Carnaxide, Lisbon District
  - Hospital Garcia de Orta, Almada
  - Hospital Central Faro, Faro